CLINICAL TRIAL: NCT01213420
Title: A Prospective, Randomized Controlled, Double Blinded, Clinical Multicentre Trial of the Aruba Aloe Formula F-BC-096 in the Treatment of Split Thickness Donor Sites After Wound Closure
Brief Title: Aruba Aloe Formula F-BC-096 in the Treatment of Split Thickness Donor Site After Wound Closure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgian Foundation for Burn Injuries, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/567
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Wounds
Keywords: Donor sites after wound closure
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aloë Vera FORMULA F-BC-096 (Experimental)
  Interventions: Other: Aloë Vera FORMULA F-BC-096 for scar hydration
- Aloë Vera FORMULA F-BC-096 with modified preservative (Active Comparator)
  Interventions: Other: Aloë Vera with modified preservative for scar hydration
- Eucerin Calming cream (Active Comparator)
  Interventions: Other: Eucerin Calming cream for scar hydration
- Nivea Cream (Active Comparator)
  Interventions: Other: Nivea Cream for scar hydration

INTERVENTIONS:
Other: Nivea Cream for scar hydration — 3 applications per day during 6 months
  Arms: Nivea Cream
Other: Aloë Vera FORMULA F-BC-096 for scar hydration — 3 applications per day during 6 months.
  Arms: Aloë Vera FORMULA F-BC-096
Other: Eucerin Calming cream for scar hydration — 3 applications per day during 6 months
  Arms: Eucerin Calming cream
Other: Aloë Vera with modified preservative for scar hydration — 3 applications per day during 6 months
  Arms: Aloë Vera FORMULA F-BC-096 with modified preservative

SUMMARY:
This study is a prospective, randomized controlled, double blinded, study in a multi centre setting. Three burn centres will include 60 patients in total.

If suited for the study (= two equal donor sites) and after informed consent, patients will be observed starting the day of skin prelevation.

A coded file will be made for each patient and these files should contain the localization of both donor sites, their depth as determined by the setting of the dermatome and the treatment. Treatment for both donor sites will always be equal.

The date of wound healing of each donor site, which may only differ by a maximum of five days, will be noted. Digital photographs of the healed donor sites will be taken and the scars will be evaluated by the local researchers using the Adapted Vancouver Scar Scale prior to the start of hydration.

From that moment on one donor site will be treated with Aruba Aloe formula F-BC-096 while one of the control products will be applied to the second site. Per group of five patients per centre a different control product will be applied to the second donor site. The tubes containing these products will be colour and numerical coded. Nor the treating personnel, nor the patients will be informed which colour tubes contain the control products and which contain the Aruba Aloe formula F-BC-096. If it is necessary to apply pressure garments for one donor site, the garments will be applied for both sites.

Follow-Ups will be performed on one, three and six months after wound closure. Objective methods will be used during these follow-ups to evaluate elasticity and colour of the scar, this by using the Dermalab, the Cutometer®, the Derma Spectrometer and the Mexameter®. The evaporation, permeability and hydration of the scar will be measured by using the Tewameter® and the Corneometer®. The Reviscometer® will measure the direction of collagen and elastin. The Adapted Vancouver Scar Scale will be used as a subjective method. Also different scales for evaluation of donor site pain, patient satisfaction, product comfort, itching etc. have to be completed by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have two similar donor sites regarding location, depth and wound treatment.
* Healing time of both donor sites may differ by 5 days maximum.
* Patient compliance with therapy in relation to the protocol is necessary. In case of paediatric patients this depends on the collaboration of the parents.
* For the two donor sites to be compared, the entire after-treatment concerning pressure garments or eventual silicone sheets must be equal for both donor sites. Pressure garments and/or silicone sheets are used only in case of burn wounds within the same location.
* Patients must be available for regular and necessary follow-up (up to 6 months post healing).
* Possibility to finish all measurements during follow-up visits.
* Written authorisation of the patient, family or parents is required.

Exclusion Criteria:

* Donor sites are not similar (not identical in: depth, wound treatment, healing time).
* The patient has a known allergy to Aloe Vera and/or to preservatives in cosmetic products.
* The patient is not able to follow the complete treatment schedule.
* The patient has any condition(s) that seriously compromises the patient's ability to complete this study.
* The occurrence of a traumatic wound over the healed donor site (e.g. abrasion, skin tear, …)
* The patient wishes to terminate the study.
* No informed consent before start of the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
improvement in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators | after 6 months of scar hydration
  * The adapted Vancouver Scar Scale (1, 3 and 6 months after wound closure)
  * Measurement of the Trans Epidermal Water Loss with the Tewameter (1, 3 and 6 months after wound closure)
  * Measurement of the hydration of the stratum corneum with the Corneometer (1, 3 and 6 months after wound closure)

SECONDARY OUTCOMES:
improvement of overall scar quality in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators: | after 6 months of scar hydration
improvement of overall product satisfaction in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators | after 6 months of scar hydration
improvement of scar colour in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators | after 6 months of scar hydration
improvement of scar elasticity in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators | after 6 months of scar hydration
improvement of collagen and elastin direction in patients treated with Aruba Aloe Formula F-BC-096 compared to patients treated with the three comparators | after 6 months of scar hydration

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital Ghent, Belgium
Locations (3):
- Belgium (3):
  - Hospital Network Antwerp, Antwerp
  - University Hospital Ghent, Ghent
  - Military Hospital, Neder-Over-Heembeek

REFERENCES:
- See also: website University Hospital Ghent, Belgium — http://www.uzgent.be